CLINICAL TRIAL: NCT00334685
Title: [S,S]-Reboxetine Add-On Trial: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center Trial Of [S,S]-Reboxetine In Patients With Postherpetic Neuralgia (PHN) Concomitantly Treated With Pregabalin.
Brief Title: [S,S]-Reboxetine Add-On Trial
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Data Monitoring Committee terminated the study on the basis of futility (insufficient clinical response).
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061021
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- [S,S]-Reboxetine + Pregabalin (Experimental)
  Interventions: Drug: [S,S]-Reboxetine + Pregabalin
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: [S,S]-Reboxetine + Pregabalin — [S,S]-Reboxetine oral, tablet 2, 4 or 6 mg per day for 10 weeks Pregabalin oral, capsule, 75, 150, 300 or 600 mg per day for 14 weeks
  Arms: [S,S]-Reboxetine + Pregabalin
Drug: Pregabalin — Pregabalin oral, capsule, 75, 150, 300 or 600 mg per day for 14 weeks
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to determine the effectiveness of adjunctive treatment of pregabalin with [S,S]-Reboxetine against pregabalin monotherapy in patients with PHN

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after the healing of shingles skin rash
* Patients at screening must have a score >/=40 mm on the pain visual analogue scale

Exclusion Criteria:

* Patients with significant renal and hepatic impairment
* Patients with other severe pain, that may impair the self-assessment of the pain due to shingles
* Patients with clinically abnormal electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2006-08-22 (Actual); Primary Completion 2007-10-04 (Actual); Study Completion 2007-10-11 (Actual)

PRIMARY OUTCOMES:
The numerical pain intensity rating scale is used to assess pain and a change from baseline in pain score for week 10 will be calculated | Week 10

SECONDARY OUTCOMES:
The mean endpoint (week 10) sleep interference score change from baseline | Week 10
Analysis of the Medical Outcomes Study Sleep Scale | Week 10
Analysis of the Patient Global Impression of Change | Week 10
Analysis of the Neuropathic Pain Symptom Inventory | Week 10

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (75):
- United States (7):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, North Dartmouth, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Kettering, Ohio
- Pfizer Investigational Site, Vienna, Austria
- Canada (14):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Langley, British Columbia
  - Pfizer Investigational Site, Greater Sudbury, Ontario
  - Pfizer Investigational Site, Hawkesbury, Ontario
  - Pfizer Investigational Site, North Bay, Ontario
  - Pfizer Investigational Site, Val Caron, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Saint Romuald, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
  - Pfizer Investigational Site, Sasktatoon, Saskatchewan
- Czechia (2):
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Pilsen
- Germany (9):
  - Pfizer Investigational Site, Erbach im Odenwald
  - Pfizer Investigational Site, Hattingen
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Katzhütte
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Münster
  - Pfizer Investigational Site, Wiesbaden
- Italy (3):
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Perugia
- Pfizer Investigational Site, Riga, Latvia
- Netherlands (2):
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Utrecht
- Norway (5):
  - Pfizer Investigational Site, Bekkestua
  - Pfizer Investigational Site, Lierskogen
  - Pfizer Investigational Site, Oslo
  - Pfizer Investigational Site, Sandnes
  - Pfizer Investigational Site, Trondheim
- Poland (2):
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Poznan
- Russia (2):
  - Pfizer Investigational Site, Saint Petersburg
  - Pfizer Investigational Site, Yaroslavl
- Spain (6):
  - Pfizer Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Pfizer Investigational Site, Cadiz
  - Pfizer Investigational Site, Granada
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia
- Sweden (5):
  - Pfizer Investigational Site, Eksjö
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Skellefteå
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site, Zurich, Switzerland
- Ukraine (7):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kharkiv
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Odesa
  - Pfizer Investigational Site, Simferopol
  - Pfizer Investigational Site, Uzhhorod
- United Kingdom (8):
  - Pfizer Investigational Site, Portsmouth, Hampshire
  - Pfizer Investigational Site, London, UK
  - Pfizer Investigational Site, Birmingham, West Midlands
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Plymouth
  - Pfizer Investigational Site, York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061021&StudyName=%5BS%2CS%5D-Reboxetine%20Add-On%20Trial